CLINICAL TRIAL: NCT06670027
Title: The Effects of Using Auditory Stimulation Methods on Cardiac Patients' Clinical Outcomes
Brief Title: The Effects of Use of Auditory Stimulation Methods on Cardiac Patients' Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Auditory stimulation
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-06

CONDITIONS: Chest Pain; Anxiety; Sleep
MeSH Terms: conditions — Chest Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Group A will receive a family voice message and Group B will be received nature sound
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family voice (Experimental): The patient receives family voice from significant member
  Interventions: Other: Family voice
- Nature sound (Active Comparator): Patient receives nature sounds such as waves sound, river streams, waterfalls, and walking in the forest
  Interventions: Other: Nature sound

INTERVENTIONS:
Other: Family voice — Group A receives the family voice
  Arms: Family voice
Other: Nature sound — Group B receives the nature sound.
  Arms: Nature sound

SUMMARY:
This study will be used to compare the effects of two auditory stimulation methods on improving vital signs parameters, reducing the severity of chest pain, and improving the sleep quality of cardiac patients.

DETAILED DESCRIPTION:
This study aims to To evaluate the relative efficacy of two auditory stimulation techniques in enhancing cardiac patients' vital sign assessments.

* This study aims to examine two auditory stimulations for their ability to alleviate chest pain in patients with heart conditions.
* The goal of this study is to evaluate two audio stimulations for their potential to help heart patients have a better night's rest.

This research made use of two different therapies including audio stimulation. Group A used familiar auditory stimulus, which was a spoken message, and group B used sounds of nature.

Patients with preexisting cardiac conditions who were admitted to a predetermined critical care unit and who subsequently intended to have percutaneous coronary artery intervention (PCI)

ELIGIBILITY:
Inclusion Criteria:

* adult (aged≥18 years).
* diagnosed with cardiac disease.
* patient with hemodynamic stability
* consciousness and ability to communicate.

Exclusion Criteria:

* patients unable to comply with study interventions
* patients with cognitive impairment
* patients with severe unstable cardiac condition
* having a history of hearing loss or the use of a hearing aid.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
sleep quality | three days after intervention
  sleep quality used Richards-Campbell Sleep Questionnaire (RCSQ). it consisted of five items score from zero mean poor pattern and 100 mean good
severity of chest pain | three days after intervention
  Visual analogue scale consisted of score from 0 to 10 zero mean no pain and 10 mean high pain
level of anxiety and depression | three days after intervention
  The hospital Anxiety and Depression (HAD) questionnaire consisted of 14 questions 7 for anxiety and 7 for depression score score 0-7 mean normal; score 8-10 mean mild; score 11-15, mean moderate; and score 16-21, mean severely

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of nursing Damanhour university, Damanhūr, Egypt